CLINICAL TRIAL: NCT00005804
Title: Treatment of Patients With Hematological Malignancies Using Marrow Transplantation From Unrelated Donors Incompatible for One HLA Locus Antigen
Brief Title: Bone Marrow Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1467.00; FHCRC-1467.00; NCI-H00-0054; CDR0000067780 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-06-02; First posted 2003-08-28 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous/Nonmalignant Condition; Small Intestine Cancer
Keywords: monoclonal gammopathy of undetermined significance; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; Burkitt lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; small intestine lymphoma; childhood immunoblastic large cell lymphoma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; recurrent/refractory childhood Hodgkin lymphoma; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; primary systemic amyloidosis; intraocular lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Recurrence; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage cancer cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of bone marrow transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence of graft-versus-host disease (GVHD) grades III and IV in patients with hematologic malignancies treated with bone marrow transplantation (BMT) using donors with 1 HLA-A or B non-cross-reactive group mismatch vs control patients previously treated with BMT using donors with 1 HLA-A or B cross-reactive group (CREG) mismatch.
* Compare the incidence of GVHD grades III and IV in patients with hematologic malignancies treated with BMT using donors with 1 HLA-A or B CREG mismatch vs control patients previously treated with BMT using matched donors.
* Determine the relevance of HLA-DRB1 or DQB1 allele mismatching in BMT using donors matched for HLA-A, B, and C.

OUTLINE: Beginning at least 3 weeks after completion of cytoreductive combination chemotherapy, patients under age 18 undergo total body irradiation (TBI) twice a day on days -7 to -4. Patients age 18 and over undergo TBI twice a day on days -6 to -4. All patients then receive cyclophosphamide IV daily on days -3 and -2. Males with acute lymphocytic leukemia, high-grade lymphoma, intermediate-grade lymphoma, or marrow or CNS involvement receive radiotherapy boost to the testes. On day 0, patients receive infusion of bone marrow from unrelated donors with 1 of the following: 1 HLA-A or B non-cross-reactive group mismatch; 1 HLA-A or B cross-reactive group mismatch; or an HLA-A, B, and C match with an HLA-DRB1 or DQB1 mismatch.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven hematologic malignancy of 1 of the following types:

  * Chronic myelogenous leukemia (CML) in chronic, accelerated, or blast* phase
  * Acute leukemia with high-risk features at diagnosis such as:

    * Philadelphia chromosome-positive acute lymphocytic leukemia**
    * Acute myeloid leukemia with high-risk cytogenetics such as inv (3), t(3;3) del(5q), -5, del(7q), -7, +8, +11, abnormal 12p, del(20q), -20, or complex abnormalities**
  * Acute leukemia with failure after one course of induction chemotherapy
  * Acute leukemia in first relapse* or second remission
  * High-risk lymphoblastic lymphoma in first remission
  * Non-Hodgkin's lymphoma, Hodgkin's disease, or other malignant lymphoproliferative disease after first remission, if an autologous transplantation is not indicated
  * Myelodysplastic or myeloproliferative syndromes ineligible for Protocol FHCRC-179 NOTE: * For patients with acute leukemia in relapse or CML in blast crisis, the search for an unrelated donor begins only if: High probability that the patient's medical condition will remain stable for the 3 to 6-month period needed to find a donorAn attempt at remission induction has been undertaken Referring physician and patient accept possibility that search for donor will be canceled if patient's condition worsens

NOTE: ** For newly diagnosed patients with high-risk acute leukemia, early referral is encouraged so that an unrelated donor search may begin immediately

* Availability of an unrelated donor with:

  * 1 HLA-A or B non-cross-reactive group (non-CREG) mismatch (except in CML in chronic phase or myelodysplastic syndrome) OR
  * 1 HLA-A or B CREG mismatch OR
  * An HLA-A, B, and C match with an HLA-DRB1 or DQB1 mismatch (no double mismatch) if 1 of the above 2 donor types unavailable

    * No more than 1 HLA-A, B, and C mismatch
* No availability of an HLA-identical sibling or haploidentical relative incompatible for 0 or 1 HLA-A or B locus of the nonshared haplotypes

  * For patients with diagnosis other than CML in chronic phase, 1 HLA-DR locus-incompatible related donor has priority over an HLA compatible or class IA or B CREG locus antigen-incompatible unrelated donor
* No severe aplastic anemia
* No leukoencephalopathy

PATIENT CHARACTERISTICS:

Age:

* Under 51
* Eligible for transplantation until age 52 if the donor is identified prior to patient's 51st birthday

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* No severe hepatic disease, including acute hepatitis

Renal:

* Creatinine less than 2 times normal

Cardiovascular:

* No cardiac insufficiency requiring treatment
* No symptomatic coronary artery disease

Pulmonary:

* No severe hypoxemia (i.e., PO2 less than 70 mm Hg) with decreased DLCO (i.e., DLCO less than 70% predicted) OR
* No mild hypoxemia (i.e., PO2 less than 80 mm Hg) with severely decreased DLCO (i.e., DLCO less than 60% predicted)
* No pulmonary fibrosis

Other:

* No other nonmalignant disease that would severely limit life expectancy
* HIV negative
* No contraindication to total body irradiation (TBI)
* Patients excluded from this study because of contraindication to TBI may be treated on protocol FHCRC-739

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy greater than 3,000 cGy to whole brain
* At least 6 months since prior involved-field radiotherapy greater than 1,500 cGy to chest or abdomen

Surgery:

* Not specified

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-10; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Anasetti, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States